CLINICAL TRIAL: NCT01175577
Title: Evaluating the Effects of Mixed-Carotenoids on Biomarkers of Endothelial Dysfunction
Brief Title: Feeding the Rainbow to Investigate Endothelial Dysfunction
Acronym: FRIED
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Bastyr University (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Ryan David Bradley, Research Assistant Professor, Bastyr University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: SP
Record Dates: First submitted 2010-08-03; First posted 2010-08-05 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Dietary Modification; Cardiovascular Disease
Keywords: mixed carotenes
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Supplement 1 (Active Comparator)
  Interventions: Dietary Supplement: Chlorophyll complex, Standard Process
- Supplement 2 (Active Comparator)
  Interventions: Dietary Supplement: Betatene, sold as "Full Spectrum Carotenoid Complex"
- Food-based Intervention (Active Comparator)
  Interventions: Other: Small carotenoid-rich meals
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Chlorophyll complex, Standard Process — One capsule, twice daily with meals for 28 days
  Arms: Supplement 1
Dietary Supplement: Betatene, sold as "Full Spectrum Carotenoid Complex" — One capsule per day with meals for 28 days
  Arms: Supplement 2
Other: Small carotenoid-rich meals — Single carotenoid-enriched soup or salad serving eaten daily
  Arms: Food-based Intervention
Other: Placebo — Safflower oil-filled capsules, one twice daily with meals
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to compare the change in blood carotene concentration between a food-based versus nutritional supplement-based intervention. This study will randomize up to 60 healthy volunteers to receive either carotenoid-enriched food; natural, mixed carotenoid supplementation; chlorophyll complex or placebo supplementation. Blood carotene levels will be measured before and after 28 days of supplementation. Preliminary data will also be collected on several biomarkers associated with vascular inflammation and endothelial dysfunction. These biomarkers will be measured before and during a fast food control meal at the beginning and end of the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18-65
* in good health by the absence of exclusion criteria on standardized medical history interview
* willingness to be randomized
* willingness to complete multiple blood draws following fast food consumption on two occasions over 28 days

Exclusion Criteria:

* children <18 years
* current use of carotenoid supplements (not including typical multivitamins containing beta-carotene)
* current use of polyphenol supplements including green tea, resveratrol, pine bark extract, cocoa, and/or grape skin extract
* current use of aspirin, statins or regular (>2 per week) use of NSAID medications
* current smoking or past smoking greater than 3 packs total or currently living with a smoker
* excessive alcohol intake (> 3 drinks per day) or history of alcoholism
* known exposure to asbestos
* autoimmune disease
* hemachromatosis
* history of gallbladder disease including gall stones or gall bladder removal
* pre-diabetes, metabolic syndrome or diabetes (1 or 2)
* established cardiovascular disease (arrhythmia, heart failure, hypertension treatment or untreated stage II hypertension (≥160/90; stage II technically diastolic ≥100mmHg, will maintain diastolic cutoff of 90mmHg), past MI or stroke)
* renal or liver disease (viral hepatitis, non-alcoholic steatohepatitis "fatty liver")
* acute infection except viral colds
* residual injury/pain/limitation from trauma
* chronic musculoskeletal disorders including osteoarthritis requiring pain medications
* psychiatric disorders that would impair completion of research tasks
* allergies to supplied foods
* anyone on a medically-prescribed diet
* >3.5 servings fruits/veggies per day
* inability to consume entire study Control meal w/in specified timeline (30 minutes)
* current pregnancy or breast feeding
* refusal to participate in blood draws following the control meal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change in serum carotenoid fraction concentrations between study arms | Following 28 day intervention

SECONDARY OUTCOMES:
Change in oxidized LDL lipoproteins (oxLDL) | Following 28 day intervention
Change in serum gamma-glutamyl transferase (GGT) | Following 28 day intervention
Change in urinary isoprostanes | Following 28 day intervention
Change in serum antioxidant capacity (ORAC) | Following 28 day intervention
Change in lipid profile (LDL, HDL, triglycerides) | Following 28 day intervention
Change in C-reactive protein (CRP) | Following 28 day intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ryan D Bradley, ND, MPH, Principal Investigator — Bastyr University
Locations (2):
- United States (2):
  - Bastyr University Clinical Research Center, Kenmore, Washington
  - University of Washington Clinical Research Center, Seattle, Washington